CLINICAL TRIAL: NCT05299398
Title: Prevention of Postpartum Depression: A Pilot Placebo-controlled Trial of Trazodone
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was pivoted to be a randomized control trial of trazodone versus quetiapine, under a new NTC identification number (study protocol number 125638).
Sponsor: Verinder Sharma (Other)
Responsible Party: Sponsor-Investigator, Verinder Sharma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 120394
Record Dates: First submitted 2021-12-30; First posted 2022-03-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Postpartum Depression
Keywords: Postpartum depression; Trazodone; Prevention
MeSH Terms: conditions — Depression, Postpartum | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trazodone (Experimental): Trazodone once daily for 24 weeks.
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator): Placebo once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trazodone — Trazodone capsule once daily
  Arms: Trazodone
Drug: Placebo — Placebo capsule once daily
  Arms: Placebo

SUMMARY:
Postpartum depression is a serious illness that affects approximately 17% of women who have recently given birth. Untreated depression appears to have negative effects for both the mother and her baby. Postpartum depression is quite common among women with a history of depression. Sleeplessness is a common concern during pregnancy and after delivery, and it can also trigger depression in women with a history of depression. Antidepressants are the most commonly recommended drugs for prevention of postpartum depression; however, there is limited research to understand the effectiveness of the medications in preventing postpartum depression. Trazodone is a weak antidepressant, but it is commonly prescribed for sleeplessness due to physical or psychiatric disorders. We are planning a study to find out whether trazodone in a low dose is more effective than a sugar pill in preventing postpartum depression among women with histories of depression. We expect the results of our study will make it easier for healthcare providers to select the right medication for women who are at risk of developing depression after delivery and thus improve the mental health of mothers and well-being of their babies.

ELIGIBILITY:
Inclusion Criteria:

Healthy outpatients with a history of Major depressive disorder who are currently not on any psychotropic medications and who:

1. are 18- 45 years old,
2. are pregnant with gestation of 28-34 weeks,
3. have been in full remission of depression for > 2 months (as per Diagnostic and Statistical Manual-5),
4. are able to communicate in English,
5. are capable of providing informed consent,
6. are planning to deliver at Victoria Hospital in London Ontario, and
7. live in London and the surrounding area, will be enrolled.

Exclusion Criteria:

1. current psychiatric disorder other than generalized anxiety,
2. use of psychotropic medication over the previous 2 months,
3. history of bipolar disorder or psychosis,
4. high risk for suicide (actively suicidal or a score of ≥ 3 on item #3 on the Hamilton Depression Rating Scale-17 item [HDRS]),
5. currently receiving psychotherapy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-17 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Major depressive episode | 27 weeks
  Participants having a score of >7 on the Hamilton Depression Rating Scale (Max 52) will be assessed using the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders- 5 (SCID-5) to establish recurrence of an major depressive episode. A higher score indicates recurrence of an MDE

SECONDARY OUTCOMES:
Time to occurrence of Major Depressive Episode (MDE) | 27 weeks
  The time from childbirth until they develop MDE
Hamilton Depression Rating Scale | 24 weeks
  The change in Hamilton Depression Rating Scale and Scale from baseline to 24 weeks to measure change in depressive symptoms. The score ranges from 0-53 where a higher score is a worse outcome.
Edinburgh Postnatal Depression | 24 weeks
  The change in Edinburgh Postnatal Depression Scale from baseline to 24 weeks to measure the change in depressive symptoms. The scores range from 0 to 30 with 30 indicating more depression symptoms.
Blood pressure | 27 weeks
  The systolic and diastolic blood pressure will be measured in mmHG.
Pulse | 27 weeks
  Pulse will be measured in Beats per minute
Body weight | 27 weeks
  Body weight will be measured in kilograms
Side effects | 27 weeks
  Side effects of Trazodone will be measured by the Frequency, Intensity, Burden of Side Effects Rating (FIBSER) scale
Maternal Functioning | 27 weeks
  Maternal Functioning will be measured by Barkin Index of Maternal Functioning. The sum of the scores is calculated, ranging from 0 to 120. Where a score of 120 means perfect functioning. The different between the scores scores will be looked at and a more positive score (8 week score is greater than baseline score) is a better outcome.
Development of mania symptoms | 27 weeks
  Mania symptoms will be measured by the Young Mania Rating Scale. here are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others. The score ranges from 0 to 60 where 60 indicates a worse outcome.
Pill count | 27 weeks
  Adherence to intervention
Retention rate | 27 weeks
  The following criteria will be used to determine the success of the study: enrollment of 1 participant every 2 weeks, and recruitment of at least 60% of all patients considered eligible to participate in the study
Complete blood count (CBC) | 27 weeks
  The CBC is a blood test to check the overall health of the participant
Thyroid Stimulating Hormone test | 27 weeks
  a blood test that measures Thyroid Stimulating Hormone measured in the units mIU/L
Electrocardiogram QT Interval | 27 weeks
  test that checks the QT interval of the heart. This will let us know if the participants have heart abnormalities or if the medication has made changes to the heart of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Verinder Sharma, MB, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Parkwood Institute Mental Health Care Building, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No